CLINICAL TRIAL: NCT00757731
Title: A European Phase III, Multicentre, Double-blind, Randomised, Monotherapy, 12-month Study of Milnacipran for the Treatment of the Fibromyalgia Syndrome
Brief Title: FMS European Long-Term Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F02207 GE 304
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Minalcipran 100 mg (Experimental)
  Interventions: Drug: milnacipran; Drug: Placebo
- Minalcipran 150 mg (Experimental)
  Interventions: Drug: milnacipran; Drug: Placebo
- Minalcipran 200 mg (Experimental)
  Interventions: Drug: milnacipran; Drug: Placebo

INTERVENTIONS:
Drug: milnacipran — hard capsule
Drug: Placebo — hard capsule

SUMMARY:
Investigation of the long-term (12 months) efficacy and safety of milnacipran used in the treatment of fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patient who completed the 3-month F02207 GE 302 study
* patient with a diagnosis of fibromyalgia according to the 1990 ACR criteria at entry of F02207 GE 302 study

Exclusion Criteria:

* known hypersensitivity to milnacipran
* major depressive episode
* significant risk of suicide
* generalised anxiety disorder
* substance abuse
* clinically significant cardiac disease
* pulmonary dysfunction
* active liver disease
* renal impairment
* autoimmune disease
* current systemic infection
* epileptic
* active cancer
* severe sleep apnoea
* active peptic ulcer
* inflammatory bowel disease
* unstable endocrine disease
* (for men) prostatic enlargement or other genito-urinary disorders
* (for women) pregnancy or breastfeeding

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To assess the long-term safety of milnacipran used for the treatment of FMS at doses of 100 mg, 150 mg and 200 mg daily | 12 months

SECONDARY OUTCOMES:
To investigate the long-term efficacy (including the durability of efficacy) of milnacipran in treating fibromyalgia over 12 months of exposure at doses of 100 mg, 150 mg and 200 mg daily | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime C BRANCO, MD, Principal Investigator — HOSPITAL EGAS MONIZ, Lisboa, Portugal
Locations (10):
- Rheumatology Ambulance, Pardubice, Czechia
- Kuopion Oma Laakari Oy, Kuopio, Finland
- Hopital Hotel Dieu, Paris, France
- KKSK KLINIKUM DER UNIVERSITAET ZU KOELN - Anaesthesiology and Intensive Care, Cologne, Germany
- Ospedale Luigi Sacco, Milan, Italy
- Center For Clinical Studies, Lillehamer, Norway
- Hospital Egas Moniz, Lisbon, Portugal
- Dr I CANTACUZINO CLINICAL HOSPITAL, Bucharest, Romania
- Hospital de La Esperanza, Barcelona, Spain
- Gottfriesclinic Ab, Mölndal, Sweden

REFERENCES:
- [Derived] Branco JC, Cherin P, Montagne A, Bouroubi A; Multinational Coordinator Study Group. Longterm therapeutic response to milnacipran treatment for fibromyalgia. A European 1-year extension study following a 3-month study. J Rheumatol. 2011 Jul;38(7):1403-12. doi: 10.3899/jrheum.101025. Epub 2011 Apr 1. PMID 21459941